CLINICAL TRIAL: NCT04370717
Title: Chronic Pain Management During a Pandemic: Will Telemedicine Replace In-person Consultation
Brief Title: Chronic Pain Management During a Pandemic
Status: Completed | Type: Observational
Sponsor: Unika Medical Centre (Network)
Responsible Party: Principal Investigator, Michael Gofeld, Principal Investigator, Unika Medical Centre
Other Study IDs: Telehealth_01
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
Keywords: chronic pain, telehealth
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: telehealth consultation — A telehealth consultation will be scheduled and conducted without modifications from the routine clinic protocol. The case report will include ICD-10 code and plan of care.
  After one week, patients will receive an electronic satisfaction survey. An in-person follow-up and/or procedural visit will be subsequently scheduled. During this visit, the same physician will complete physical examination, document the diagnosis and proceed with either the same or modified plan of care. The research coordinator will enter diagnostic and procedural codes in the case report form.
  Other Names: in-person visit

SUMMARY:
This is an open-label cohort study of chronic pain patients referred to an interdisciplinary community outpatient clinic. The aim of this study is to determine whether video consultations are non-inferior to regular consultations in diagnosing and planning subsequent interventions. The null hypothesis is that there is no difference in the International Statistical Classification of Diseases 10th edition (ICD-10) codes established via telehealth and subsequent clinic visits. The patients will complete standard health questionnaires online and undergo a structured and detailed interview to clarify the diagnosis and establish appropriate treatment. A limited telehealth physical examination based on direct observation will be conducted.

At the subsequent clinic visit, the accuracy of diagnosis and adherence to the plan of care will be evaluated.

The primary and secondary endpoints will be gathered from the electronic charts and from the recruited participants by questionnaires completed online one week after the telemedicine consultation. The diagnosis and plan of care semi-structured match will be performed during the in-person follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

all patients referred for consultation

Exclusion Criteria:

1. Not English-speakers
2. Patients who do not have any compatible telecommunication devices
3. Patients illiterate in basic telecommunication and have no one in their household to help
4. Patients unable to complete online self-assessment forms and study questionnaires
5. Patients unable to make a follow-up visit
6. Individuals with unstable pain complaints

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive community patients referred to the interdisciplinary clinic
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a matching diagnosis between telehealth and in-person consultation | 6 months

SECONDARY OUTCOMES:
Percentage of patients with a matching plan of care/recommendations between telehealth and in-person visit | 6 months
Patient satisfaction from telehealth encountered measured on 7-point Likert scale | 6 months
feasibility of telehealth visits | 6 months
  (a) percentage of patients who accepted telemedicine as an equal substitute to in-person consultation. Participants will be asked the question with possible answers "Yes" or "No", "Why Yes?" "Why No?" (b) dropout rates and causes of dropouts (medical or technical reasons) will be registered (c) participants' satisfaction with video quality and sound quality (patients will be asked if they were "satisfied" with the video quality and sound quality after telemedicine consultation; "Yes" or "No", "Why not?"), (d) technical errors with the telemedicine equipment, and (e) specialist consultation time in minutes.
cost-saving | 6 months
  Calculated cost-saving included (a) cost of travel in Canadian dollars, (b) estimated loss of income (<3.5 hours=a half day's salary, >3.5 hours spent on travel and consultation=one day's salary), (c) travelling distance in kilometres and travelling time in hours as estimated by Google Maps.

CONTACTS AND LOCATIONS:
Locations (1):
- Silver Centre for Pain Care, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website of the participating clinic — https://silverpaincare.com/